CLINICAL TRIAL: NCT04470609
Title: A Randomized, Double-blind, Placebo-controlled, Phase Ib/IIb Trial of an Inactivated SARS-CoV-2 Vaccine in Healthy People Aged ⩾60 Years
Brief Title: Safety and Immunogenicity Study of an Inactivated SARS-CoV-2 Vaccine for Preventing Against COVID-19 in People Aged ⩾60 Years
Status: Completed | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: Institute of Medical Biology, Chinese Academy of Medical Sciences (Other)
Collaborators: West China Second University Hospital (Other); Yunnan Center for Disease Control and Prevention (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Prevention
Other Study IDs: 20200402
Record Dates: First submitted 2020-07-13; First posted 2020-07-14 (Actual); Last update posted 2023-10-11 (Actual); Status verified 2023-10

CONDITIONS: COVID-19
MeSH Terms: conditions — COVID-19 | interventions — Appointments and Schedules

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (4):
- Low dosage vaccine on a 0- and 28-day schedule (Experimental): Two doses of low dosage Inactivated SARS-CoV-2 Vaccine at the vaccination schedule of day 0, 28
  Interventions: Biological: Low dosage Inactivated SARS-CoV-2 Vaccine on a 0- and 28-day schedule
- Medium dosage vaccine on a 0- and 28-day schedule (Experimental): Two doses of medium dosage Inactivated SARS-CoV-2 Vaccine at the vaccination schedule of day 0, 28
  Interventions: Biological: Medium dosage Inactivated SARS-CoV-2 Vaccine on a 0- and 28-day schedule
- High dosage vaccine on a 0- and 28-day schedule (Experimental): Two doses of high dosage Inactivated SARS-CoV-2 Vaccine at the vaccination schedule of day 0, 28
  Interventions: Biological: High dosage Inactivated SARS-CoV-2 Vaccine on a 0- and 28-day schedule
- Placebo on a 0- and 28-day schedule (Placebo Comparator): Two doses of placebo at the vaccination schedule of day 0, 28
  Interventions: Biological: Placebo on a 0- and 28-day schedule

INTERVENTIONS:
Biological: Low dosage Inactivated SARS-CoV-2 Vaccine on a 0- and 28-day schedule — Two doses of low dosage(50U/0.5ml) Inactivated SARS-CoV-2 Vaccine at the vaccination schedule of day 0,28
  Arms: Low dosage vaccine on a 0- and 28-day schedule
Biological: Medium dosage Inactivated SARS-CoV-2 Vaccine on a 0- and 28-day schedule — Two doses of medium dosage(100U/0.5ml) Inactivated SARS-CoV-2 Vaccine at the vaccination schedule of day 0,28
  Arms: Medium dosage vaccine on a 0- and 28-day schedule
Biological: High dosage Inactivated SARS-CoV-2 Vaccine on a 0- and 28-day schedule — Two doses of high dosage(150U/0.5ml) Inactivated SARS-CoV-2 Vaccine at the vaccination schedule of day 0,28
  Arms: High dosage vaccine on a 0- and 28-day schedule
Biological: Placebo on a 0- and 28-day schedule — Two doses of placebo at the vaccination schedule of day 0,28
  Arms: Placebo on a 0- and 28-day schedule

SUMMARY:
This study is a randomized, double-blinded, and placebo-controlled phase Ib/IIb clinical trial of the Inactivated SARS-CoV-2 Vaccine to evaluate the safety and immunogenicity of the vaccine in healthy people aged ⩾60 Years.

DETAILED DESCRIPTION:
This phase Ib/IIb trial is designed to evaluate the safety and immunogenicity of different doses of the Inactivated SARS-CoV-2 Vaccine based upon the randomized, double-blind and placebo-controlled principle. A total of 471 subjects aged ⩾60 years will be enrolled in the study, of which 96 and 375 will be enrolled for phase Ib and phase Ⅱb,respectively. The enrolled subjects in phase Ib receive two doses of low-, medium-, or high-dose of experimental vaccines or placebo at an interval of 28 days, while the enrolled subjects in Phase Ⅱb receive two doses of medium, high-dose experimental vaccines or placebo at an interval of 28 days.

ELIGIBILITY:
Inclusion Criteria:

* Phase Ib:

  1. Healthy people aged ⩾60 years (including boundary values), both men and women.
  2. Proven legal identity.
  3. Participants should understand the contents of the informed consent form, the vaccine in this trial, voluntarily sign the informed consent form, and be capable of using thermometers, scales, and filling in diary cards and contact cards as required.
  4. Participants should be able to communicate well with investigators, understand and comply with the requirements of this trial.
  5. Axillary temperature ≤37.0 ℃.
* Phase IIb:

  1. Healthy people aged ⩾60 years (including boundary values), both men and women.
  2. Proven legal identity.
  3. Participants should understand the contents of the informed consent form, the vaccine in this trial, voluntarily sign the informed consent form, and be capable of using thermometers, scales, and filling in diary cards and contact cards as required.
  4. Participants should be able to communicate well with investigators, understand and comply with the requirements of this trial.
  5. Axillary temperature ≤37.0 ℃.

Exclusion Criteria:

* Phase Ib:

  1. Contraindications for vaccination.
  2. History of allergy to vaccines or drugs.
  3. Immunization with any vaccine within 1 month.
  4. Diseases that cannot be controlled by drugs, such as hypertension, diabetes, asthma, etc.
  5. Those who developed acute disease within 2 weeks, or had symptoms of fever or upper respiratory tract infection within 7 days.
  6. Those who have a hereditary bleeding tendency or coagulation dysfunction, or a history of thrombosis or bleeding disorders.
  7. Those who cannot tolerate venipuncture, or have a history of halo needles or halo blood.
  8. For any reason, the spleen was removed partially or completely.
  9. Those who have undergone surgery within 3 months before signing the informed consent, or those who plan to perform surgery during the trial or within 3 months after the end of the trial (including cosmetic surgery, dental and oral surgery).
  10. Those who donated or lost blood (≥200 mL) in the past 3 months, who received blood transfusion or use of blood products, or who planned blood donation during the trial.
  11. Receipt of other investigational or unregistered products (drugs, vaccines, biological product or devices) in the past 3 months, or plan to use other investigational or unregistered products during the study.
  12. Receipt of immunosuppressive therapy within 6 months before signing the informed consent form, such as long-term systemic glucocorticoid therapy (with systemic glucocorticoid therapy for more than 2 weeks within 6 months, such as prednisone or similar drugs) ), but local administration (such as ointment, eye drops, inhalation, or nasal spray) is allowed. The local administration should not exceed the dosage recommended in the instructions or have any signs of systemic exposure.
  13. Those who have took soft drugs (such as marijuana) within 3 months before signing the informed consent form or took hard drugs (such as: cocaine, phencyclidine, etc.) within 1 year before the trial.
  14. Those who smoked more than 5 cigarettes per day within 3 months before signing the informed consent form.
  15. The weekly drinking volume is greater than 14 units within 3 months before signing the informed consent form (1 unit alcohol approximately equal to 360 mL beer or 45 mL spirits with 40% alcohol content or 150 mL wine).
  16. The comprehensive physical examination does not meet the health standards, mainly including: (1) Those with abnormal vital signs with clinical significance. (2) BMI<18 kg/m^2 or> 30 kg/m^2. (3) Abnormal laboratory examination with clinical significance. (4) Those who tested positive for human immunodeficiency virus (HIV) antibody, hepatitis B surface antigen, hepatitis B e antigen, hepatitis C virus antibody, or Treponema pallidum antibody (tp-trust).
  17. Women who have a positive pregnancy test, or men who have a birth plan or plan to donate sperm from the screening to 12 months after the second vaccination.
  18. Positive in drug abuse screening during the screening period (Morphine, Methamphetamine, Ketamine, MDMA and Tetrahydrocannabinolic acid).
  19. Positive in alcohol breath test during the screening period.
  20. Positive in SARS-CoV-2 nucleic acid screening or antibodies (IgG or IgM) screening.
  21. History of severe acute respiratory syndrome (SARS) or Middle East respiratory syndrome (MERS) or other coronavirus infection (HCoV-229E, HCoV-OC43, HCoV-NL63, HCoV-HKU1).
  22. History of contact with confirmed or suspected cases infected with SARS-CoV-2 within 1 month.
  23. Any other situations judged by investigators as not suitable for participating in this study.
* Phase IIb:

  1. Contraindications for vaccination.
  2. History of allergy to vaccines or drugs.
  3. Immunization with any vaccine within 1 month.
  4. Diseases that cannot be controlled by drugs, such as hypertension, diabetes, asthma, etc.
  5. Those who developed acute disease within 2 weeks, or had symptoms of fever or upper respiratory tract infection within 7 days.
  6. Those who have a hereditary bleeding tendency or coagulation dysfunction, or a history of thrombosis or bleeding disorders.
  7. For any reason, the spleen was removed partially or completely.
  8. Those who have undergone surgery within 3 months before signing the informed consent, or those who plan to perform surgery during the trial or within 3 months after the end of the trial (including cosmetic surgery, dental and oral surgery).
  9. Those who donated or lost blood (≥200 mL) in the past 3 months, who received blood transfusion or use of blood products, or who planned blood donation during the trial.
  10. Receipt of other investigational or unregistered products (drugs, vaccines, biological product or devices) in the past 3 months, or plan to use other investigational or unregistered products during the study.
  11. Receipt of immunosuppressive therapy within 6 months before signing the informed consent form, such as long-term systemic glucocorticoid therapy (with systemic glucocorticoid therapy for more than 2 weeks within 6 months, such as prednisone or similar drugs) ), but local administration (such as ointment, eye drops, inhalation, or nasal spray) is allowed. The local administration should not exceed the dosage recommended in the instructions or have any signs of systemic exposure.
  12. Women who have a positive pregnancy test, or men who have a birth plan or plan to donate sperm from the screening to 12 months after the second vaccination.
  13. History of severe acute respiratory syndrome (SARS) or Middle East respiratory syndrome (MERS) or other coronavirus infection (HCoV-229E, HCoV-OC43, HCoV-NL63, HCoV-HKU1).
  14. History of contact with confirmed or suspected cases infected with SARS-CoV-2 within 1 month.
  15. The comprehensive physical examination does not meet the health standards, mainly including: (1) Those with abnormal vital signs (Pulse <55 beats per minute or> 100 beats per minute at rest, Systolic blood pressure ≥140mmHg or Diastolic blood pressure ≥90mmHg, breathing> 20 beats per minute or <12 beats per minute). (2) Those who tested positive for human immunodeficiency virus (HIV) antibody, hepatitis B surface antigen, hepatitis B e antigen, hepatitis C virus antibody, or Treponema pallidum antibody (tp-trust).
  16. Positive in SARS-CoV-2 nucleic acid screening or antibodies (IgG or IgM) screening.
  17. Any other situations judged by investigators as not suitable for participating in this study.

Min Age: 60 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 471 (Actual)
Dates: Start 2020-07-10 (Actual); Primary Completion 2020-10-30 (Actual); Study Completion 2021-10-27 (Actual)

PRIMARY OUTCOMES:
Adverse reactions/events rate | 7 days after vaccination
  Occurence of adverse reactions/events after vaccination
Adverse reactions/events rate | 28 days after vaccination
  Occurence of adverse reactions/events after vaccination
Seroconversion rate of Neutralizing antibodies against SARS-CoV-2 Phase IIb | 28 days after vaccination
  Seroconversion rate of neutralizing antibodies against SARS-CoV-2 in serum for Phase IIb with vaccination schedule of day 0, 28
Seroconversion rate of IgG antibodies against SARS-CoV-2 Phase IIb | 28 days after vaccination
  Seroconversion rate of IgG antibodies against SARS-CoV-2 tested by ELISA in serum for Phase IIb with vaccination schedule of day 0, 28

SECONDARY OUTCOMES:
Serious adverse events | 12 months after the second vaccination
  Occurence of Serious adverse events after vaccination
Seroconversion rate of Neutralizing antibodies against SARS-CoV-2 Phase Ib | 28 days after the second vaccination
  Seroconversion rate of neutralizing antibodies against SARS-CoV-2 in serum for Phase Ib with vaccination schedule of day 0, 28
Seroconversion rate of IgG antibodies against SARS-CoV-2 Phase Ib | 28 days after the second vaccination
  Seroconversion rate of IgG antibodies against SARS-CoV-2 tested by ELISA in serum for Phase Ib with vaccination schedule of day 0, 28
Level of Neutralizing antibodies against SARS-CoV-2 Phase Ib | 7 and 28 days after the second vaccination
  Level of neutralizing antibodies against SARS-CoV-2 in serum for Phase Ib with vaccination schedule of day 0, 28
Level of IgG antibodies against SARS-CoV-2 Phase Ib | 7 and 28 days after the second vaccination
  Level of IgG antibodies against SARS-CoV-2 tested by ELISA in serum for Phase Ib with vaccination schedule of day 0, 28
Level of Neutralizing antibodies against SARS-CoV-2 Phase IIb | 28 days after the second vaccination
  Level of neutralizing antibodies against SARS-CoV-2 in serum for Phase IIb with vaccination schedule of day 0, 28
Level of IgG antibodies against SARS-CoV-2 Phase IIb | 28 days after the second vaccination
  Level of IgG antibodies against SARS-CoV-2 tested by ELISA in serum for Phase IIb with vaccination schedule of day 0, 28

OTHER OUTCOMES:
Level of IgM antibodies against SARS-CoV-2 Phase Ib | 7 and 28 days after the second vaccination
  Level of IgM antibodies against SARS-CoV-2 tested by ELISA in serum for Phase Ib with vaccination schedule of day 0, 28
Level of Neutralizing antibodies against SARS-CoV-2 Phase Ib | 3, 6, 9 and 12 months after the second vaccination
  Level of neutralizing antibodies against SARS-CoV-2 in serum for Phase Ib with vaccination schedule of day 0, 28
Level of IgG antibodies against SARS-CoV-2 Phase Ib | 3, 6, 9 and 12 months after the second vaccination
  Level of IgG antibodies against SARS-CoV-2 tested by ELISA in serum for Phase Ib with vaccination schedule of day 0, 28
Cellular immune responses Phase Ib | 7 and 28 days after the second vaccination
  Cellular immune responses (CD4+, CD8+, Th1, Th2, IFN-γ, TNFα, IL-2, IL-6) will be measured for Phase Ib with vaccination schedule of day 0, 28
Level of IgM antibodies against SARS-CoV-2 Phase IIb | 28 days after the second vaccination
  Level of IgM antibodies against SARS-CoV-2 tested by ELISA in serum for Phase IIb with vaccination schedule of day 0, 28
Level of anti-N protein antibodies Phase IIb | 28 days after the second vaccination
  Level of anti-N protein antibodies for Phase IIb with vaccination schedule of day 0, 28
Level of Neutralizing antibodies against SARS-CoV-2 Phase IIb | 6 and 12 months after the second vaccination
  Level of neutralizing antibodies against SARS-CoV-2 in serum for Phase IIb with vaccination schedule of day 0, 28
Level of IgG antibodies against SARS-CoV-2 Phase IIb | 6 and 12 months after the second vaccination
  Level of IgG antibodies against SARS-CoV-2 tested by ELISA in serum for Phase IIb with vaccination schedule of day 0, 28
Cellular immune responses Phase IIb | 28 days after the second vaccination
  Cellular immune responses (CD4+, CD8+, Th1, Th2, IFN-γ, TNFα, IL-2, IL-6) will be measured for Phase IIb with vaccination schedule of day 0, 28

CONTACTS AND LOCATIONS:
Overall Officials: Qin Yu, Principal Investigator — West China Second University Hospital; Xiaoqiang Liu, Principal Investigator — Yunnan Center for Disease Control and Prevention
Locations (1):
- West China Second University Hospital, Sichuan University / West China women's and children's Hospital, Chengdu, Sichuan, China